CLINICAL TRIAL: NCT02862262
Title: A Multi-Site Clinical Evaluation of the ARIES Bordetella Assay in Symptomatic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Luminex Molecular Diagnostics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: LMA-BRD-01-CS-001
Record Dates: First submitted 2016-07-12; First posted 2016-08-11 (Estimated); Last update posted 2018-10-04 (Actual); Status verified 2018-10

CONDITIONS: Bordetella Infections; Bordetella Pertussis Infection; Bordetella Parapertussis Infection
MeSH Terms: conditions — Bordetella Infections; Whooping Cough

STUDY DESIGN:
Intervention Model Description: The study is comprised of three arms:
  Arm 1: Blinded, Prospective Arm Primary arm comprised of prospectively collected, de-identified, left-over nasopharyngeal swab specimens.
  Arm 2: Blinded, Pre-selected Arm Because both B. pertussis and B. parapertussis exhibited low prevalence rates in the prospective study cohort, the prospective sample set was supplemented with banked (pre-selected) positive specimens collected at selected sites.
  Arm 3: Contrived Specimens Because the number of B. parapertussis positive clinical specimens tested in Arm 1 and Arm 2 of the study was insufficient for accurate estimate of positive percent agreement (PPA) for this target, fifty (50) contrived specimens spiked with relevant B. parapertussis strains at different levels were also prepared. The analyte concentrations covered clinically relevant titers.
Masking Description: All eligible specimens (de-identified remnants) enrolled are tested using both the investigational device as well as the reference method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Blinded, Prospective Arm (1) (Experimental): Clinical performance of the ARIES Bordetella Assay for the detection of B. pertussis and B. parapertussis will be evaluated in prospectively collected, de-identified, left-over, clinical specimens.
  Interventions: Device: ARIES Bordetella Assay
- Blinded, Pre-selected Arm (2) (Experimental): In the event that an insufficient number of positive specimens are acquired for B. pertussis / B. parapertussis in Arm 1, clinical performance of the ARIES Bordetella Assay will be tested using banked, pre-selected, positive clinical specimens.
  Interventions: Device: ARIES Bordetella Assay
- Blinded, Contrived Arm (3) (Experimental): Contrived specimens will be tested using the ARIES Bordetella Assay to evaluate detection of B. parapertussis in the event that an insufficient number of positive specimens are acquired in Arm 2.
  Interventions: Device: ARIES Bordetella Assay

INTERVENTIONS:
Device: ARIES Bordetella Assay

SUMMARY:
A three-arm, multi-site clinical evaluation of the ARIES Bordetella Assay for the detection and identification of Bordetella pertussis (B. pertussis) and Bordetella parapertussis (B. parapertussis) nucleic acids in prospectively collected, de-identified, left-over clinical specimens; banked, pre-selected clinical specimens; and contrived specimens.

DETAILED DESCRIPTION:
The ARIES Bordetella Assay is a real-time polymerase chain reaction (PCR) based qualitative in vitro diagnostic test for the direct detection and identification of Bordetella pertussis (B. pertussis) and Bordetella parapertussis (B. parapertussis) nucleic acid in nasopharyngeal swabs (NPS) specimens obtained from individuals suspected of having a respiratory tract infection attributable to B. pertussis or B. parapertussis.

Clinical nasopharyngeal swab specimens collected using nasopharyngeal swab in transport media will be processed according to the routine procedure followed at the clinical collection site and as ordered by the referring physician. The leftover specimen will be blinded and assigned a unique clinical study specimen number. In order to preserve the confidentiality of subjects, the following procedures will be implemented at each site:

* Clinical specimens will be individually numbered by an honest broker who is not involved in investigational testing so that the identity of the subject may not be readily ascertained by the investigator, investigational testing staff, or study Sponsor.
* Available clinical information accompanying the specimens will be provided in such a way that it does not make the specimen source identifiable to the investigator or any other individuals associated with investigational testing, including the Sponsor.
* No personal identifier (protected health information) will be included on the case report form (CRF) so that the confidentiality of each subject is protected.

Multiple aliquots of each left-over specimen will be generated. One aliquot of each specimen will be shipped to a laboratory where the reference method (two validated real-time PCR methods for each, B. pertussis and B. parapertussis) will be performed. A second aliquot of each specimen will be used by the clinical sites for ARIES Bordetella Assay testing. Additional aliquots of each specimen will be stored frozen (-65 to -95°C) at the clinical sites and sent separately on dry ice to the Sponsor upon Sponsor's request.

The prospective data set will be supplemented with banked, pre-selected clinical specimens and contrived specimens that tested positive by a comparator method for B. pertussis and B. parapertussis. If contrived specimens are required, these specimens will be prepared then blinded, aliquoted, randomized and frozen (-65 to -95°C) until distributed to the clinical testing sites by the Sponsor.

The clinical data will be automatically generated from the ARIES System software. The system will report the specimen as B. pertussis and B. parapertussis positive (Co-infection), B. pertussis positive, B. parapertussis positive, B. pertussis and B. parapertussis negative or Invalid. Invalid results will be retested and both the original data and the retest data will be reported. The clinical data will be compared to the reference data and recorded in the clinical study reports.

ELIGIBILITY:
Inclusion Criteria:

1. The specimen is a nasopharyngeal swab collected using a cleared nasopharyngeal swab and transport medium.
2. The specimen is from an adult or pediatric, male or female subject who is either hospitalized, admitted to a hospital emergency department, visiting an outpatient clinica or resident of a long term care facility.
3. The specimen is from a patient for whom a requisition has been made for B. pertussis and/or B. parapertussis testing.
4. The specimen is from a patient exhibiting clinical signs and symptoms of respiratory tract infection consistent with B. pertussis or B. parapertussis.
5. The specimen was received in good condition (no leakage or drying of the specimen).
6. The specimen contains a minimum volume of 1000 μL.

Exclusion Criteria:

1. The specimen is not a nasopharyngeal swab collected using a cleared nasopharyngeal swab and transport medium.
2. The specimen was not properly collected, transported, processed or stored according to the instructions provided by the Sponsor in Section 10 below.
3. The specimen volume is <1000 μL.
4. Any specimen that was not tested per the complete testing algorithm provided by the Sponsor.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1052 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11-14 (Actual)

PRIMARY OUTCOMES:
Specificity and sensitivity of the ARIES Bordetella Assay in patients suspected of having respiratory infection attributable to B. pertussis or B. parapertussis. | 5 months
  Estimates of positive percent agreement and negative percent agreement for each target will be calculated based on a two-by-two table (reference method result vs. result from ARIES Bordetella Assay) for each target. In addition, 95% two sided confidence intervals will be provided. Positive agreement and negative agreement values will be provided for the entire prospective data set.

SECONDARY OUTCOMES:
Clinical performance of the ARIES Bordetella Assay per clinical site. | 5 months
  Positive agreement and negative agreement values will be provided for each clinical site.
Clinical performance of the ARIES Bordetella Assay per age group. | 5 months
  Positive agreement and negative agreement values will be provided for pediatric vs. adult patients.
Clinical performance of the ARIES Bordetella Assay per patient sub-population. | 5 months
  Positive agreement and negative agreement values will be provided for each patient sub population (e.g., immuno-competent vs. immuno-compromised patients, and hospitalized vs. outpatient vs. long-term care facility).

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Dunn, Study Director — Luminex Molecular Diagnostics; Timothy S Uphoff, PhD, Principal Investigator — Marshfield Labs; Stephen Young, PhD, Principal Investigator — Tricore Reference Lab; Ryan Relich, PhD, Principal Investigator — IU Health Pathology Laboratory; Ted E Schutzbank, PhD, Principal Investigator — St. John Hospital & Medical Center; Amy L Leber, PhD, Principal Investigator — Nationwide Children's Hospital Laboratory
Locations (6):
- United States (5):
  - Indiana University Health, Indianapolis, Indiana
  - St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Tricore, Albuquerque, New Mexico
  - Nationwide Children's Hospital Laboratory, Columbus, Ohio
  - Marshfield Labs, Marshfield, Wisconsin
- Luminex Molecular Diagnostics, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Relich RF, Leber A, Young S, Schutzbank T, Dunn R, Farhang J, Uphoff TS. Multicenter Clinical Evaluation of the Automated Aries Bordetella Assay. J Clin Microbiol. 2019 Jan 30;57(2):e01471-18. doi: 10.1128/JCM.01471-18. Print 2019 Feb. PMID 30518543